CLINICAL TRIAL: NCT04350697
Title: Comparison Between Ministernotomy and Minithoracotomy for Aortic Surgery
Brief Title: Mini-invasive Approaches to Aortic Surgery
Acronym: MSvsMT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Florence (Other)
Collaborators: Prof Sandro Gelsomino (Unknown); Prof Edvin Prifti (Unknown); Prof Guido Sani (Unknown); Dr Aleksander Dokollari (Unknown)
Responsible Party: Principal Investigator, Massimo Bonacchi, Professor, University of Florence
Other Study IDs: MSvsMT
Record Dates: First submitted 2020-04-07; First posted 2020-04-17 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2020-04

CONDITIONS: Surgery; Surgical Injury; Surgical Procedure, Unspecified; Surgical Incision; Aortic Surgery
Keywords: miniinvasive surgery; aortic surgery; minithoracotomy; ministernotomy; outcomes; surgical complications
MeSH Terms: conditions — Intraoperative Complications; Surgical Wound

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mini-Sternotomy: Patients underwent aortic surgery by Mini-Sternotomy
  Interventions: Procedure: Aortic Surgery
- Mini-Thoracotomy: Patients underwent aortic surgery by Mini-Thoracotomy
  Interventions: Procedure: Aortic Surgery

INTERVENTIONS:
Procedure: Aortic Surgery — Surgery for aortic and/or aortic valve diseases

SUMMARY:
There are many different types of mini-invasive approaches to aortic surgery. Ministernotomy and anterior right minithoracotomy are the two main techniques applied for minimally invasive aortic valve replacement, but if one of them is superior in terms of patient outcomes it is not still clear. Therefore, the aim of this study is to compare the immediate and long-term outcomes of these two techniques.

ELIGIBILITY:
Inclusion Criteria:

- Indication for Aortic and/or Aortic Valve surgery

Exclusion Criteria:

- none

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery for Aortic and/or Aortic Valve by miniinvasive approaches (ministernotomy or minithoracotomy)
Sampling Method: Non-Probability Sample
Enrollment: 2425 (Estimated)
Dates: Start 1999-01-01; Primary Completion 2021-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PO | 1 day after surgery
  Post-Operative Survival

SECONDARY OUTCOMES:
EO | 1 month after surgery
  Early Outcome (Survival)
MO | 5 years after surgery
  Mid-term Outcome (Survival)
LO | 10 years after surgery
  Late Outcome (Survival)
VLO | 20 years after surgery
  Very-Late Outcome (Survival)

CONTACTS AND LOCATIONS:
Locations (1):
- Massimo Bonacchi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bonacchi M, Dokollari A, Parise O, Sani G, Prifti E, Bisleri G, Gelsomino S. Ministernotomy compared with right anterior minithoracotomy for aortic valve surgery. J Thorac Cardiovasc Surg. 2023 Mar;165(3):1022-1032.e2. doi: 10.1016/j.jtcvs.2021.03.125. Epub 2021 Apr 23. PMID 33994208